CLINICAL TRIAL: NCT03175211
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Subcutaneous Doses of BI 456906 in Healthy Male Subjects (Single-blind, Partially Randomised, Placebo-controlled Parallel Group Design)
Brief Title: Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BI 456906 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1404-0001; 2017-000295-29 (EudraCT Number)
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-02

CONDITIONS: Healthy
MeSH Terms: interventions — BI 456906

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 456906 (Experimental)
  Interventions: Drug: BI 456906
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 456906 — single dose
  Arms: BI 456906
Drug: Placebo — single dose
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of BI 456906 in healthy subjects following single rising doses.

The secondary objective is the exploration of the pharmacokinetics including dose proportionality, and pharmacodynamics (PD) of BI 456906 after single dosing

ELIGIBILITY:
Inclusion criteria

* Healthy male according to the assessment of the Investigator, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (incl.)
* Body Mass Index (BMI) of 20.0 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Further exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
[N (%)] of subjects with drug-related adverse events. | Up to 672 hours

SECONDARY OUTCOMES:
AUC0-168 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 168h) | up to 168 hours
Cmax (maximum measured concentration of the analyte in plasma) | up to 672 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

REFERENCES:
- [Derived] Jungnik A, Arrubla Martinez J, Plum-Morschel L, Kapitza C, Lamers D, Thamer C, Scholch C, Desch M, Hennige AM. Phase I studies of the safety, tolerability, pharmacokinetics and pharmacodynamics of the dual glucagon receptor/glucagon-like peptide-1 receptor agonist BI 456906. Diabetes Obes Metab. 2023 Apr;25(4):1011-1023. doi: 10.1111/dom.14948. Epub 2023 Jan 30. PMID 36527386